CLINICAL TRIAL: NCT05422794
Title: A Phase 1b Trial of ZEN003694 (ZEN-3694) With Pembrolizumab and Nab-Paclitaxel in Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: Testing the Addition of Anti-Cancer Drug, ZEN003694 (ZEN-3694) and PD-1 Inhibitor (Pembrolizumab), to Standard Chemotherapy (Nab-Paclitaxel) Treatment in Patients With Advanced Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-04956; NCI-2022-04956 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DFHCC #22-589; 10525 (Other: Dana-Farber - Harvard Cancer Center LAO); 10525 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Triple-Negative Breast Carcinoma; Metastatic Triple-Negative Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (ZEN003694, nab-paclitaxel, pembrolizumab) (Experimental): Patients receive ZEN003694 PO QD on days 1-21, nab-paclitaxel IV over 30 minutes on day 1, 8, and 15, and pembrolizumab IV over 30 minutes every 21 days of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity with a maximum of 35 doses of pembrolizumab administered. Patients also undergo CT or MRI scan and collection of blood samples throughout the trial.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Nab-paclitaxel; Biological: Pembrolizumab
- Dose Expansion (ZEN003694, nab-paclitaxel, pembrolizumab) (Experimental): Patients receive ZEN003694 PO QD on days 1-7 prior to combination therapy. Patients then receive ZEN003694 PO QD on days 1-21, nab-paclitaxel IV over 30 minutes on days 1, 8, and 15, and pembrolizumab IV over 30 minutes every 21 days of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity with a maximum of 35 doses of pembrolizumab administered. Patients also undergo biopsies on study, and CT or MRI scans and collection of blood samples throughout the trial.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Nab-paclitaxel; Biological: Pembrolizumab

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Dose Expansion (ZEN003694, nab-paclitaxel, pembrolizumab)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase Ib trial tests the safety and tolerability of ZEN003694 in combination with an immunotherapy drug called pembrolizumab and the usual chemotherapy approach with nab-paclitaxel for the treatment of patients with triple negative-negative breast cancer that has spread to other parts of the body (advanced). Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of paclitaxel which may have fewer side effects and work better than other forms of paclitaxel. Immunotherapy with monoclonal antibodies, such as pembrolizumab may help the body's immune system attach the cancer and may interfere with the ability of tumor cells to grow and spread. ZEN003694 is an inhibitor of a family of proteins called the bromodomain and extra-terminal (BET). It may prevent the growth of tumor cells that over produce BET protein. Combination therapy with ZEN003694 pembrolizumab immunotherapy and nab-paclitaxel chemotherapy may help shrink or stabilize cancer for longer than chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of BET bromodomain inhibitor ZEN-3694 (ZEN003694) used in combination with pembrolizumab and nab-paclitaxel in patients with locally advanced or metastatic triple negative-negative breast cancer (TNBC).

II. Evaluate the safety and tolerability of ZEN003694 used in combination with pembrolizumab and nab-paclitaxel in patients with locally advanced or metastatic TNBC.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. Confirm the recommended phase 2 dose (RP2D) from the trial by assessing the totality of the evidence (i.e., safety, tolerability, pharmacokinetic, and activity data) from this trial to select an optimal dosage(s) for future trials with registrational intent.

III. Evaluate the pharmacokinetic (PK) profile of the combination of ZEN003694, pembrolizumab and nab-paclitaxel.

IV. Determine the preliminary efficacy of the combination of ZEN003694, pembrolizumab and nab-paclitaxel, as assessed by overall response rate (ORR), progression-free survival (PFS), overall survival (OS), duration of response (DoR) and time to objective response (TTOR), utilizing Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, in patients with locally advanced or metastatic TNBC.

V. Quantify changes in PD-L1 pre- and post-exposure to BET bromodomain inhibitor (BBDI) and determine correlations that occur with response to the triplet combination.

VI. Quantify cytotoxic T cell populations, T cell activation, checkpoint expression, and angiogenesis and determine if location or absolute number of CD8+ T cells pre- and post-exposure to BBDI is predictive of response to immunotherapy with the triplet combination.

VII. Determine whether differential gene expression of immune-activating and immunosuppressive pathways occurs with exposure to single-agent BBDI and/or to the triplet combination of BBDI, PD-1 inhibition and taxane-based chemotherapy, and whether these changes correlate with response or resistance to treatment.

EXPLORATORY OBJECTIVES:

I. Explore potential biomarker indicators of response and resistance to the triplet combination in tumor tissue, blood, and stool samples.

OUTLINE: This is a dose-escalation study of ZEN003694 in combination with fixed-dose pembrolizumab and nab-paclitaxel, followed by a dose-expansion study.

DOSE ESCALATION: Patients receive ZEN003694 orally (PO) once daily (QD) on days 1-21, nab-paclitaxel intravenously (IV) over 30 minutes on day 1, 8, and 15, and pembrolizumab IV over 30 minutes every 21 days of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity with a maximum of 35 doses of pembrolizumab administered. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) scan and collection of blood samples throughout the trial.

DOSE EXPANSION: Patients receive ZEN003694 PO QD on days 1-7 prior to combination therapy. Patients then receive ZEN003694 PO QD on days 1-21, nab-paclitaxel IV over 30 minutes on days 1, 8, and 15, and pembrolizumab IV over 30 minutes every 21 days of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity with a maximum of 35 doses of pembrolizumab administered. Patients also undergo biopsies on study, and CT or MRI scans and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up for 30 days after the last dose of study medication and then every 6 months for a maximum of 3 years or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed diagnosis of TNBC based on standard criteria for the disease:

  * Estrogen receptor (ER) and progesterone receptor (PR) < 10% by immunohistochemistry (IHC), and HER2-negative (per current American Society of Clinical Oncology [ASCO]/College of American Pathologists [CAP] guidelines)
  * If there is more than one histological result available, the most recent sample with ER, PR and HER2 results will be considered for inclusion
  * Patients who have not had ER, PR and HER2 testing and thus, ER, PR and HER2 status is unknown, are not eligible
  * Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation
* Participants must have disease that is unresectable locally advanced or metastatic
* DOSE ESCALATION COHORT: Known PD-L1 status is not required prior to study enrollment. Central PD-L1 testing (on archival tumor tissue) will occur retrospectively
* DOSE ESCALATION COHORT: Any number of prior lines of therapy are allowed in the metastatic setting. Prior immune checkpoint inhibitor allowed in any setting
* DOSE ESCALATION COHORT: Evaluable or measurable disease per RECIST 1.1 criteria
* DOSE EXPANSION COHORT: PD-L1 status must be negative. Standard local testing with any PD-L1 antibody that has been validated in a Clinical Laboratory Improvement Act (CLIA)- certified environment will be acceptable for including patients on trial. Primary or metastatic samples may be tested for PD-L1 status. Central confirmation will occur retrospectively. For patients in whom a baseline research tumor tissue biopsy is not performed (e.g. site of disease is not safely accessible), archival tissue should be provided for central confirmatory PD-L1 testing
* DOSE EXPANSION COHORT: 0-1 prior lines of systemic therapy in the metastatic setting
* DOSE EXPANSION COHORT: Participants must have measurable disease per RECIST 1.1 criteria
* DOSE EXPANSION COHORT: Participants must have disease that is amenable to biopsy as judged by the treating investigator and must be willing to undergo pre- and on-treatment tumor biopsies, if safely accessible
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of ZEN003694 (ZEN-3694) in combination with nab-paclitaxel and pembrolizumab (MK-3475) in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (or =< 2.0 x ULN in patients with documented Gilbert's Syndrome)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3.0 x institutional ULN or ≤ 5.0 x institutional ULN for participants with documented liver metastases
* Serum or plasma creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min (based on the calculated chronic kidney disease epidemiology (CKD-EPI) glomerular filtration rate estimation
* International normalized ratio (INR) or prothrombin time (PT): =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT): =< 1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial as long as their anti-retroviral therapy does not have the potential for drug-drug interactions as judged by the treating investigator
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with history of treated central nervous system (CNS) metastases are eligible, provided they meet the following criteria:

  * Disease outside the CNS is present
  * Recovery from acute toxicity associated with the treatment to =< Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 or baseline (with the exception of alopecia), with no requirement for escalating doses of corticosteroids over the past 7 days
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer are allowed
* Patients should be New York Heart Association Functional Classification of class 2B or better
* Peripheral neuropathy grade =< 1
* Ability to swallow and retain oral medications
* Participants may not have had cytotoxic chemotherapy, immunotherapy, major surgery (other than diagnostic surgery, dental surgery or stenting), or other investigational therapy within 3 weeks prior to entering the study
* Participants may not have had radiotherapy within 1 week prior to entering the study. Patients may not have had > 25% of their bone marrow radiated. Stereotactic radiosurgery (SRS) within 1 week prior to entering the study will be allowed
* Participants may not have received tyrosine kinase inhibitors (TKIs) or small molecules within 5 half-lives or 2 weeks (whichever is shorter) of study entry
* Patients who have experienced adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) must have recovered, with the exception of alopecia or as otherwise specified in the eligibility criteria
* The effects of the combination of ZEN003694 (ZEN-3694) and MK-3475 on the developing human fetus are unknown. For this reason and because BETi and PD-1 blocking agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after study completion. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of ZEN003694 (ZEN-3694), MK-3475 and nab-Paclitaxel administration. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to registration. Childbearing potential is defined as: participants who have not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus)
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZEN003694 (ZEN-3694), nab-paclitaxel, or pembrolizumab
* Patients with uncontrolled intercurrent illness
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Any gastrointestinal (GI) disorder that may affect absorption of oral medications in the opinion of the treating investigator, such as malabsorption syndrome or major bowel or stomach resection
* Pregnant women are excluded from this study because ZEN003694 (a BETi agent) and MK-3475 have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZEN003694 (ZEN-3694), breastfeeding should be discontinued if the mother is treated with ZEN003694 (ZEN-3694). These potential risks may also apply to MK-3475 and nab-paclitaxel
* Patients who have previously received ZEN003694 (ZEN-3694) or who have been treated with an investigational BET inhibitor
* DOSE EXPANSION COHORT: Prior exposure to immune checkpoint inhibitors in the metastatic setting. PD-1 or PD-L1 inhibitors in the neo-/adjuvant setting are allowed if at least 12 months have elapsed since the end of adjuvant systemic treatment to development of metastatic disease
* DOSE EXPANSION COHORT: Prior exposure to taxane-based therapy in the metastatic setting. Taxane in the neo-/adjuvant setting is allowed if at least 12 months have elapsed since the end of adjuvant systemic treatment to development of metastatic disease
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Strong inhibitors or inducers of CYP3A4 must be discontinued at least 7 days prior to the first dose of ZEN003694 (ZEN-3694). Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients receiving any medications or substances that are Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
* Patients who have had a bone-targeted radionuclide within 6 weeks of the first dose of ZEN003694 (ZEN-3694)
* Myocardial infarction or unstable angina within 6 months prior to the first dose of ZEN003694 (ZEN-3694)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI)
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has a known history of active tuberculosis (TB)
* Has received a live vaccine within 30 days of planned treatment start. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacille Calmette-Guerin (BCG), and typhoid vaccine. Seasonal flu vaccines that do not contain live virus are permitted. Coronavirus disease-2019 (COVID-19) vaccines received within the last 30 days are also permitted
* Participants with known or suspected extensive bone marrow infiltration per radiographic assessment, laboratory assessment, or bone marrow sampling (e.g., aspiration or biopsy), determined to be clinically significant by the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ZEN003694 (ZEN-3694) used in combination with pembrolizumab and nab-paclitaxel | Up to 28 days from start of treatment
  A Bayesian optimal interval design will be used to identify the MTD.
Recommended phase 2 dose (RP2D) of ZEN003694 (ZEN-3694) used in combination with pembrolizumab and nab-paclitaxel | Up to 28 days from start of treatment
  Will be for adverse events consistent with a dose-limiting toxicity definition.
Incidence of adverse events | Up to 3 years from treatment start date
  Toxicity will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0. Toxicities will be summarized by maximum grade and by treatment dose level. Incidence rate of each toxicity will be reported with 95% exact confidence intervals.

SECONDARY OUTCOMES:
Pharmacokinetics profile of the combination of ZEN003694 (ZEN-3694), pembrolizumab and nab-paclitaxel | Pre-dose & 2 hours (h) post-dose on cycle 0 day 1 (C0D1), C2D15, C4D1, & C6D8; pre-dose & 0.5h post-dose on C1D1; pre-dose & 0.5, 1, 2, 4, 6, 8 & 24h post-dose on C1D15
  Given the potential for interactions via CYP3A4, the pharmacokinetics of both ZEN003694 (ZEN-3694) and paclitaxel are assessed to confirm whether a clinically relevant drug-drug interaction occurs. Plasma concentration-time curves will be analyzed by noncompartmental methods using routines supplied in the Phoenix WinNonlin. For pembrolizumab, the primary assessment will be individual baseline pembrolizumab clearance as a continuous variable in uni-variate and multi-variate Cox proportional hazards models for progression free survival (PFS).
Recommended phase 2 dose (RP2D) | Up to 3 years
  Will confirm the RP2D from the trial by assessing the totality of the evidence (i.e., safety, tolerability, pharmacokinetic, and activity data) from this trial to select an optimal dosage(s) for future trials with registrational intent. Toxicity will be graded according to NCI CTCAE, Version 5.0. Toxicities will be summarized by maximum grade and by treatment dose level. Incidence rate of each toxicity will be reported with 95% exact confidence intervals.
Overall response rate | From start of the treatment until disease progression/ recurrence, or for up to 3 years
  Radiographic response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and will be graded as complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). All patients (dose escalation, triple negative breast cancer [TNBC] unselected by PD-L1 status; dose expansion, TNBC PD-L1-negative) who receive at least one dose of study treatment will be included in the efficacy analyses.
PFS | From the time of study enrollment until the identification of disease progression or death, or for up to 3 years
  Radiographic response will be assessed by RECIST 1.1 criteria and will be graded as CR, PR, SD, and PD. Subjects without disease progression or death at the time of analysis will be censored at the date of last known alive. All patients (dose escalation, TNBC unselected by PD-L1 status; dose expansion, TNBC PD-L1-negative) who receive at least one dose of study treatment will be included in the efficacy analyses.
Overall survival | From the time of study enrollment until death due to any cause, or for up to 3 years
  Subjects without disease progression or death at the time of analysis will be censored at the date of last known alive. All patients (dose escalation, TNBC unselected by PD-L1 status; dose expansion, TNBC PD-L1-negative) who receive at least one dose of study treatment will be included in the efficacy analyses.
Duration of response (DoR) | Time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease, or for up to 3 years
  Radiographic response will be assessed by RECIST 1.1 criteria and will be graded as CR, PR, SD, and PD. Median DOR will be reported with ranges. All patients (dose escalation, TNBC unselected by PD-L1 status; dose expansion, TNBC PD-L1-negative) who receive at least one dose of study treatment will be included in the efficacy analyses.
Time to objective response (TTOR) | From start of treatment to the time, measurement criteria are met for CR or PR (whichever is first recorded), or for up to 3 years
  Radiographic response will be assessed by RECIST 1.1 criteria and will be graded as CR, PR, SD, and PD. Median TTOR will be reported with ranges. All patients (dose escalation, TNBC unselected by PD-L1 status; dose expansion, TNBC PD-L1-negative) who receive at least one dose of study treatment will be included in the efficacy analyses.
Changes in potential biomarkers | Baseline up to post-treatment biopsies
  Multiplex immunofluorescence (IF) will be performed on formalin-fixed paraffin-embedded sections of tumor tissue specimens to evaluate the presence, distribution and interaction of different immune cell populations utilizing validated multiplex IF panels. The integrated biomarker panel includes the following markers: pancytokeratin, CD8, PD-1, PD-L1, and CD31.

OTHER OUTCOMES:
Potential biomarker indicators of response and resistance to the triplet combination | Baseline up to on-treatment and post-treatment biopsies
  To characterize the expression of tumor markers by immunohistochemistry and/or IF, descriptive statistics and agglomerative hierarchical clustering techniques will be used to summarize the distribution and patterns of profiles observed in baseline samples. Descriptive statistics will be used to summarize the change in markers and inferences on treatment-effects will use non-parametric tests (e.g. Wilcoxon rank sum) with two-sided alpha 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Garrido-Castro, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (6):
- United States (6):
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm